CLINICAL TRIAL: NCT01054430
Title: A PHASE I, OPEN LABEL, NON-RANDOMIZED, SINGLE-DOSE, PARALLEL-COHORT, MATCHED-CONTROL STUDY TO EVALUATE THE PHARMACOKINETICS AND SAFETY OF AVANAFIL (TA-1790) IN SUBJECTS WITH HEPATIC IMPAIRMENT AND IN HEALTHY CONTROL MALE SUBJECTS
Brief Title: To Assess the Safety of Avanafil in Healthy and Hepatically Impaired Male Subjects.
Acronym: avanafil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, VP Clinical, Vivus, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA-012
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Erectile Dysfunction
Keywords: Avanafil; Hepatic; Erectile Dysfunction; Impairment
MeSH Terms: conditions — Erectile Dysfunction | interventions — avanafil

ARMS (3):
- Normal (Other): Subjects with normal hepatic function
  Interventions: Drug: avanafil
- Mild Hepatic Dysfunction (Other): Subjects with mild hepatic impairment
  Interventions: Drug: avanafil
- Moderate hepatic dysfunction (Other): Subjects with moderal hepatice impairment
  Interventions: Drug: avanafil

INTERVENTIONS:
Drug: avanafil — 200 mg avanafil tablets QD

SUMMARY:
The objective of this study is to assess the single dose pharmacokinetics of avanafil in subjects with hepatic impairment and in healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects must be 21-75 years of age; inclusive. Healthy control subjects (Cohort 1) must be medically healthy with clinically insignificant screening results and hepatically impaired subjects (Cohorts 2 and 3) must have mild or moderate hepatic impairment based on the Child-Pugh Classification.

Exclusion Criteria:

* Main exclusion criteria for healthy control subjects (Cohort 1) include history or clinical evidence of clinically relevant cardiovascular (including thromboembolic disorders), hepatic, renal, hematologic, endocrine, pulmonary, gastrointestinal, psychiatric or neurological impairment; any clinically significant laboratory abnormalities as judged by the investigatorInvestigator; systolic blood pressure < 90 or >160 mmHg; diastolic blood pressure < 50 or > 90 mmHg; allergy to or previous adverse events with PDE5 inhibitors; use of prescription or over-the-counter drugs that are known to interfere with metabolism by the cytochrome P450 3A4 enzyme within 30 days of screening; use of any investigational drug within 30 days of screening; use of any prescription or over-the-counter drugs or herbal remedies within 14 days of screening; history of alcohol or drug abuse within 18 months, history of smoking within 6 months; positive breath alcohol test; positive serology for HIV, HCV, HBsAg; blood donation or significant blood loss within 56 days of dosing; plasma donation within 7 days of dosing.

Main exclusion criteria for hepatically impaired subjects (Cohorts 2 and 3) include any significant concurrent medical condition or history of significant medical conditions other than hepatic impairment that may affect the interpretation of the data or which otherwise contraindicates participation in this study; acute exacerbation of or unstable hepatic disease, as indicated by worsening of clinical and/or laboratory signs of hepatic impairment, within the 2 weeks preceding study drug administration; history of esophageal variceal bleeding within past 6 months; history of bleeding or non-bleeding gastric varices; history of spontaneous bacterial peritonitis within the past 3 months; history of portosystemic surgical shunt; autoimmune liver disease; history of organ transplant; Wilson's disease; diagnosis of cholestatic liver disease (e.g., primary biliary cirrhosis or primary sclerosing cholangitis); history of recent symptomatic cryoglobulinemia; alcoholic hepatitis, determined clinically or by histology; initiation of any new prescription or over the counter medications within 14 days before study drug administration and hemoglobin < 9.0 g/dL, positive for AFP.

Ages: 21 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Single Dose Pharmacokinetics of avanafil | 1 day

SECONDARY OUTCOMES:
single dose safety | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Shiyin Yee, PhD, Study Director — VIVUS LLC